CLINICAL TRIAL: NCT03306940
Title: Does Bilateral Botulinum Toxin A in Patients With Hemifacial Spasm Improve Facial Symmetry Unilateral and Bilateral Injection of Botulinum Toxin A in Patients With Hemifacial Spasm? A Prospective, Randomized, Controlled Study
Brief Title: Botulinum Toxin A in the Treatment of Hemifacial Spasm
Acronym: BTATHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Lingjing Jin, professor, Tongji University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14SG21
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Hemifacial Spasm
Keywords: botulinum toxin A
MeSH Terms: conditions — Hemifacial Spasm | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unilateral injection group (Placebo Comparator): Patients of unilateral group were injected botulinum toxin type A to the affected hemiface.
  Interventions: Drug: Botulinum Toxin Type A
- bilateral injection group (Experimental): Patients of bilateral group were injected botulinum toxin type A to the affected hemiface and normal hemiface. The intervention of the bilateral group was that the normal side was injected.
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — patients were injected to the normal side with dose of 1.25 units/per site
  Other Names: Chinese botulinum toxin type A

SUMMARY:
Hemifacial spasm patients who received botulinum toxin A injection were divided into two groups. Group A received unilateral injection while group B received bilateral injection. Patients completed follow-up A researcher record facial videos and analyzed facial symmetry and completed 3 scales.

DETAILED DESCRIPTION:
Hemifacial spasm patients who received botulinum toxin A injection were divided into two groups.Patients of unilateral group were injected to the affected side and the dose of botulinum toxin A was 2.5-3.75 units/per site. Patients of bilateral group were injected to the affected side with dose of 2.5-3.75 units/per site and the normal side was injected with dose of 1.25 units/per site.

3 scales for measurement were used.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hemifacial spasm
* Scott grading III to IV
* hemifacial spasm duration of half or more years
* last botulinum toxin A application at least 3 months before the start of the study

Exclusion Criteria:

* history of facial trauma, congenital facial asymmetry, facial nerve microsurgical decompression
* bilateral hemifacial spasm
* allergies to botulinum toxin A or to any component of the drug
* previous treatment with botulinum toxin A fewer than 3 months
* the use of drugs that could interfere with neuromuscular transmission or spasm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Sunnybrook Facial Grading System | up to 6 months
  Sunnybrook Facial Grading System consists of resting symmetry, symmetry of voluntary movement and synkinesis. Total score = Symmetry of voluntary movement score - Resting symmetry score - Synkinesis score

SECONDARY OUTCOMES:
Symmetry Scale for Hemifacial Spasm | up to 6 months
  Symmetry Scale for Hemifacial Spasm consists of resting symmetry and symmetry of voluntary movement. Total score =Resting symmetry score + Symmetry of voluntary movement score
Facial Clinimetric Evaluation Scale | up to 6 months
  Facial Clinimetric Evaluation Scale consists of six parts:facial movement,facial comfort,oral function,eye comfort,lacrimal control and social function. Total score = facial movement + facial comfort + oral function + eye comfort + lacrimal control + social function.
The effective duration of botulinum toxin A | up to 6 months
  degree of amelioration in spasm and the effective duration of botulinum toxin A
Adverse events | up to 6 months
  Adverse events, including stiff face, difficulty drinking and eating, difficulty controlling parotid and so on.The onset and duration of adverse events.Whether to take intervention to ameliorate adverse events and the efficacy of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lingjing Jin, PhD, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tan NC, Chan LL, Tan EK. Hemifacial spasm and involuntary facial movements. QJM. 2002 Aug;95(8):493-500. doi: 10.1093/qjmed/95.8.493. PMID 12145388
- [Result] Fujimura T, Hotta M. The preliminary study of the relationship between facial movements and wrinkle formation. Skin Res Technol. 2012 May;18(2):219-24. doi: 10.1111/j.1600-0846.2011.00557.x. Epub 2011 Aug 25. PMID 22092807
- [Result] Isse NG. Endoscopic facial rejuvenation: endoforehead, the functional lift. Case reports. Aesthetic Plast Surg. 1994 Winter;18(1):21-9. doi: 10.1007/BF00444243. PMID 8122572
- [Result] Xiao L, Pan Y, Zhang X, Hu Y, Cai L, Nie Z, Pan L, Li B, He Y, Jin L. Facial asymmetry in patients with hemifacial spasm before and after botulinum toxin A treatment. Neurol Sci. 2016 Nov;37(11):1807-1813. doi: 10.1007/s10072-016-2670-2. Epub 2016 Jul 18. PMID 27431279
- [Result] Kim J. Contralateral botulinum toxin injection to improve facial asymmetry after acute facial paralysis. Otol Neurotol. 2013 Feb;34(2):319-24. doi: 10.1097/mao.0b013e31827c9f58. PMID 23444480
- [Result] Borodic GE, Cheney M, McKenna M. Contralateral injections of botulinum A toxin for the treatment of hemifacial spasm to achieve increased facial symmetry. Plast Reconstr Surg. 1992 Dec;90(6):972-7; discussion 978-9. PMID 1448532